CLINICAL TRIAL: NCT01387282
Title: Anamorelin HCl in the Treatment of Non-Small Cell Lung Cancer-Cachexia (NSCLC-C): A Randomized Double-Blind Placebo-Controlled Multicenter Phase III Study to Evaluate the Safety and Efficacy of Anamorelin HCl in Patients With NSCLC-C
Brief Title: Safety and Efficacy of Anamorelin HCl in Patients With Non-Small Cell Lung Cancer-Cachexia (ROMANA 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helsinn Therapeutics (U.S.), Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HT-ANAM-302
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-09

CONDITIONS: Cachexia; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Cachexia; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 100 mg QD (Active Comparator): Investigational: Anamorelin HCl; 100 mg tablets; oral administration QD for 12 weeks, at least 1 hour before the first meal of the day.
  Interventions: Drug: Anamorelin HCl
- Placebo (Placebo Comparator): Placebo tablets identical in appearance to active tablets; oral administration once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anamorelin HCl — Anamorelin HCL 100 mg will be orally administered daily at least 1 hour prior to meal
  Arms: 100 mg QD
Drug: Placebo — Placebo tablets identical in appearance to active tablets; oral administration QD for 12 weeks, at least 1 hour prior to meal before the first meal of the day.
  Arms: Placebo

SUMMARY:
The administration of Anamorelin in patients with Stage III-IV non-small cell lung cancer-cachexia (NSCLC-C) is expected to increase appetite, lean body mass, weight gain, and muscle strength.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter study to assess the safety and efficacy of Anamorelin in patients with non-small cell lung cancer-cachexia (NSCLC-C). The primary efficacy analysis will include the treatment difference in the change in lean body mass and physical function.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of unresectable Stage III or Stage IV NSCLC
* Patients may be receiving maintenance chemotherapy
* Patients planning to initiate a new chemotherapy and/or radiation therapy regimen may do so only within ± 14 days of randomization
* Patients may have completed a chemotherapy and/or radiation therapy and/or have no plan to initiate a new regimen within 12 weeks from randomization; at least 14 days must elapse from the completion of the chemotherapy and/or radiation therapy prior to randomization
* Involuntary weight loss of ≥5% body weight within 6 months prior to screening or a screening body mass index (BMI) <20 kg/m2
* Body mass index ≤30 kg/m2
* Life expectancy of >4 months at time of screening
* ECOG performance status ≤2
* Adequate hepatic function, defined as AST and ALT levels ≤5 x upper limit of normal
* Adequate renal function, defined as creatinine ≤2 x upper limit of normal, or calculated creatinine clearance >30 ml/minute
* Ability to understand and comply with the procedures for the HGS evaluation
* If a woman of childbearing potential or a fertile man, he/she must agree to use an effective form of contraception during the study and for 30 days following the last dose of study drug (an effective form of contraception is abstinence, a hormonal contraceptive, or a double-barrier method)
* Must be willing and able to give signed informed consent and, in the opinion of the Investigator, to comply with the protocol tests and procedures

Exclusion Criteria:

* Other forms of lung cancer (e.g., small cell, mesothelioma)
* Women who are pregnant or breast-feeding
* Known HIV, hepatitis (B&C), or active tuberculosis
* Had major surgery (central venous access placement and tumor biopsies are not considered major surgery) within 4 weeks prior to randomization; patients must be well recovered from acute effects of surgery prior to screening; patients should not have plans to undergo major surgical procedures during the treatment period
* Currently taking prescription medications intended to increase appetite or treat weight loss; these include, but are not limited to, testosterone, androgenic compounds, megestrol acetate, methylphenidate, and dronabinol
* Inability to readily swallow oral tablets; patients with severe gastrointestinal disease (including esophagitis, gastritis, malabsorption, or obstructive symptoms) or intractable or frequent vomiting are excluded
* Has an active, uncontrolled infection
* Has uncontrolled diabetes mellitus
* Has untreated clinically relevant hypothyroidism
* Has known or symptomatic brain metastases
* Receiving strong CYP3A4 inhibitors within 14 days of randomization
* Receiving tube feedings or parenteral nutrition (either total or partial); patients must have discontinued these treatments for at least 6 weeks prior to Day 1, and throughout the study duration
* Other clinical diagnosis, ongoing or intercurrent illness that in the Investigator's opinion would prevent the patient's participation
* Has had previous exposure to Anamorelin HCl
* Patients actively receiving a concurrent investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2011-07; Primary Completion 2013-11 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (46):
- United States (14):
  - Corona, California
  - Fountain Valley, California
  - Glendale, California
  - Washington D.C., District of Columbia
  - Baltimore, Maryland
  - Detroit, Michigan
  - Lake Success, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Sylvania, Ohio
  - West Reading, Pennsylvania
  - Charleston, South Carolina
  - Falls Church, Virginia
- Australia (4):
  - Prairiewood, New South Wales
  - East Bentleigh, Victoria
  - Parkville, Victoria
  - Adelaide
- Hungary (5):
  - Budapest
  - Nyíregyháza
  - Székesfehérvár
  - Szikszó
  - Törökbálint
- Israel (8):
  - Beersheba
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Petach Tikvah
  - Tel Aviv
  - Tel Litwinsky
  - Ẕerifin
- Poland (8):
  - Bydgoszcz
  - Grudziądz
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Szczecin
  - Warsaw
- Russia (5):
  - Krasnodar
  - Moscow
  - Novosibirsk
  - Saint Petersburg
  - Yekaterinburg
- United Kingdom (2):
  - Leicester
  - Middlesex

REFERENCES:
- [Derived] Laird BJA, Skipworth R, Bonomi PD, Fallon M, Kaasa S, Giorgino R, McMillan DC, Currow DC. Anamorelin Efficacy in Non-Small-Cell Lung Cancer Patients With Cachexia: Insights From ROMANA 1 and ROMANA 2. J Cachexia Sarcopenia Muscle. 2025 Feb;16(1):e13732. doi: 10.1002/jcsm.13732. PMID 39992021
- [Derived] Currow D, Temel JS, Abernethy A, Milanowski J, Friend J, Fearon KC. ROMANA 3: a phase 3 safety extension study of anamorelin in advanced non-small-cell lung cancer (NSCLC) patients with cachexia. Ann Oncol. 2017 Aug 1;28(8):1949-1956. doi: 10.1093/annonc/mdx192. PMID 28472437
- [Derived] Temel JS, Abernethy AP, Currow DC, Friend J, Duus EM, Yan Y, Fearon KC. Anamorelin in patients with non-small-cell lung cancer and cachexia (ROMANA 1 and ROMANA 2): results from two randomised, double-blind, phase 3 trials. Lancet Oncol. 2016 Apr;17(4):519-531. doi: 10.1016/S1470-2045(15)00558-6. Epub 2016 Feb 20. PMID 26906526
- [Derived] Salsman JM, Beaumont JL, Wortman K, Yan Y, Friend J, Cella D. Brief versions of the FACIT-fatigue and FAACT subscales for patients with non-small cell lung cancer cachexia. Support Care Cancer. 2015 May;23(5):1355-64. doi: 10.1007/s00520-014-2484-9. Epub 2014 Oct 29. PMID 25351456

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 477 patients with advanced NSCLC-C (defined as unresectable Stage III and Stage IV and a weight loss of ≥ 5% body weight within 6 months prior to screening or a screening body mass index [BMI] < 20 kg/m2) were to be randomized 2:1 to anamorelin HCl 100 mg or placebo.
Pre-assignment Details: Central randomization stratified patients by geographic region, by chemotherapy and/or radiation therapy status and by weight loss over prior 6 months.
Groups:
- Anamorelin HCl: Active drug; 100 mg tablets; oral administration QD for 12 weeks, at least 1 hour before the first meal of the day.
- Placebo: Placebo tablets identical in appearance to active tablets; oral administration QD for 12 weeks, at least 1 hour before the first meal of the day.
Period: Overall Study
Arm/Group | Anamorelin HCl | Placebo
Started | 330 | 165
ITT Population | 330 | 165
MITT Population | 268 | 136
Safety Population | 330 | 161
Completed (A patient was considered to have completed the study if the patient completed Week 12/Day 85 Visit.) | 233 | 118
Not Completed | 97 | 47
Not completed — Death | 47 | 16
Not completed — Other | 5 | 1
Not completed — Unrelated AE | 6 | 4
Not completed — Withdrawal by patient | 33 | 23
Not completed — Study drug-related AE | 2 | 2
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anamorelin HCl | Placebo | Total
Number analyzed (Participants) | 330 | 165 | 495
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 209 | 108 | 317
  >=65 years | 121 | 57 | 178
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 43 | 133
  Male | 240 | 122 | 362
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 1 | 3
  White | 326 | 162 | 488
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Poland | 133 | 70 | 203
  United Kingdom | 1 | 0 | 1
  Hungary | 72 | 36 | 108
  Australia | 14 | 8 | 22
  Israel | 8 | 5 | 13
  Russian Federation | 92 | 41 | 133
  United States | 10 | 5 | 15
Geographic region [Count of Participants; unit: Participants]
  North America | 10 | 5 | 15
  West Europe | 142 | 75 | 217
  East Europe + Russia | 164 | 77 | 241
  Australia | 14 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Lean Body Mass
Description: Change in Lean Body Mass (LBM) from baseline over 12 weeks for the ITT Population. Change from baseline over 12 weeks was defined as the average of the change from baseline at Week 6 and the change from baseline at Week 12.
Time Frame: Change in Lean Body Mass from Baseline Over 12 Weeks
Population: Intent-to-Treat Population. Some patients in the ITT population were excluded from the primary LBM/HGS analysis (i.e., multiple imputations/ranking method) if they survived to Week 12 but missed their baseline covariates including LBM, HGS, or ECOG OR had Week 6 and Week 12 outcomes that were outside the visit windows.
Measure: Median (95% Confidence Interval); unit: kg
Arm/Group | Anamorelin HCl | Placebo
Number analyzed (Participants) | 321 | 157
kg | 0.65 [0.38 to 0.91] | -0.98 [-1.49 to -0.41]
Statistical Analysis 1: Comparison: Anamorelin HCl vs Placebo; Superiority analysis; Test type: Superiority or Other; p < 0.0001, Wilcoxon rank sum test

2. Primary Outcome: Change in Handgrip Strength
Description: Change in Handgrip Strength (HGS) of the non-dominant hand from baseline over 12 weeks for the ITT Population. Change from baseline over 12 weeks was defined as the average of the change from baseline at Week 6 and the change from baseline at Week 12.
Time Frame: Change in Handgrip Strength of the Non-Dominant Hand from Baseline Over 12 Weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: kg
Arm/Group | Anamorelin HCl | Placebo
Number analyzed (Participants) | 321 | 157
kg | -1.49 [-2.06 to -0.58] | -0.95 [-1.56 to 0.04]
Statistical Analysis 1: Comparison: Anamorelin HCl vs Placebo; Superiority analysis; Test type: Superiority or Other; p = 0.6480, Wilcoxon rank sum test

3. Secondary Outcome: Change in A/CS Domain Score
Description: The Functional Assessment of Anorexia/Cachexia Treatment (FAACT) Additional Concerns Subscale (A/CS domain) is a 12-item scale that is part of the Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System. Each item is answered on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much).
  The 12-items are summed together to obtain the domain score. Note that negatively phrased questions are reverse scored so that higher scores always represent improvement/less symptom burden. The total possible score for the A/CS domain ranges from 0 (worst) to 48 (best).
Time Frame: Change in FAACT A/CS Domain Score from Baseline Over 12 Weeks
Population: Modified Intent-to-Treat Population
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Anamorelin HCl | Placebo
Number analyzed (Participants) | 268 | 136
scores on a scale | 3.48 (0.944) | 1.34 (1.032)
Statistical Analysis 1: Comparison: Anamorelin HCl vs Placebo; Superiority analysis; Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis

4. Secondary Outcome: Change in FACIT-F Fatigue Domain Score
Description: The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) fatigue domain is a 13-item scale that is part of the Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System. Each item is answered on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much).
  The 13-items are summed together to obtain the domain score. Note that negatively phrased questions are reverse scored so that higher scores always represent improvement/less symptom burden. The total possible score for the FACIT-F fatigue domain ranges from 0 (worst) to 52 (best).
Time Frame: Change in FACIT-F Fatigue Domain Score from Baseline Over 12 Weeks
Population: Modified Intent-to-Treat Population
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Anamorelin HCl | Placebo
Number analyzed (Participants) | 268 | 136
scores on a scale | 1.37 (1.169) | 1.23 (1.293)
Statistical Analysis 1: Comparison: Anamorelin HCl vs Placebo; Superiority analysis; Test type: Superiority or Other; p = 0.8637, Mixed Models Analysis

5. Secondary Outcome: Change in Body Weight
Description: Change in body weight (BW) from baseline overall (i.e., over 12 weeks) for the MITT Population.
Time Frame: Change in Body Weight from Baseline Over 12 Weeks
Population: Modified Intent-to-Treat Population
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Anamorelin HCl | Placebo
Number analyzed (Participants) | 268 | 136
kg | 0.95 (0.386) | -0.57 (0.438)
Statistical Analysis 1: Comparison: Anamorelin HCl vs Placebo; Superiority analysis; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse events that occurred during the clinical trial, commenced with the first dose of study drug through the 28 day post-treatment follow-up visit.
Description: Adverse events that occurred following the signature of the informed consent, but prior to the first dose of study drug were not reported as adverse events in this trial. The adverse event reporting period also ended if the patient began an alternative therapy within 28 days of the last administration of study drug. The Safety Population, defined as all randomized patients who received any study drug, was used for all safety analyses.
Arm/Group | Anamorelin HCl | Placebo
Serious Adverse Events (participants affected / at risk) | 73/330 | 27/161
Other Adverse Events (participants affected / at risk) | 156/330 | 72/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anamorelin HCl (N=330) | Placebo (N=161)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 25 (25) | 10 (10)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Epiglottic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatine increased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 1 (1) | 0 (0)
cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pulmonary haemorrhage (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 1 (1)
cerebrovasculary insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anamorelin HCl (N=330) | Placebo (N=161)
Anaemia (Blood and lymphatic system disorders) | 48 (61) | 21 (28)
Leukopenia (Blood and lymphatic system disorders) | 25 (29) | 6 (7)
Neutropenia (Blood and lymphatic system disorders) | 31 (48) | 10 (14)
Asthenia (General disorders) | 29 (30) | 16 (19)
Nausea (Gastrointestinal disorders) | 19 (20) | 13 (13)
Vomiting (Gastrointestinal disorders) | 9 (11) | 9 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 29 (35) | 14 (15)
Hyperglycaemia (Metabolism and nutrition disorders) | 23 (32) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor intends to publish the complete study results in a timely manner that is appropriate to the project. Separate publication of a portion of the study results by any PI is discouraged.